CLINICAL TRIAL: NCT06384248
Title: An Open, Single-Arm, Phase II Clinical Study Evaluating the Efficacy and Safety of LTC004 Alone in Patients With Locally Advanced or Metastatic Sarcoma Who Have Failed Standard Treatment
Brief Title: Phase II Clinical Study of LTC004 in Patients With Advanced Sarcoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Letolab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTC004-205
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Unresectable or Metastatic Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHASE 1 (Experimental): Enrollment of 10 consecutive evaluable sarcoma subjects with failure of existing standard therapy or lack of effective treatment Treated with LTC004 in Phase I
  Interventions: Drug: LTC004
- PHASE 2 (Experimental): If ≥2 subjects experience objective remission or SD lasting >12 weeks in PHASE 1, proceed to Phase II to enroll an additional 20 evaluable subjects to further evaluation of the safety and efficacy of LTC004
  Interventions: Drug: LTC004

INTERVENTIONS:
Drug: LTC004 — LTC004,45μg/kg,IV,Day 1,Q3W;

SUMMARY:
This is a phase II clinical study to evaluate the safety, tolerability and preliminary antitumor activity of LTC004 in patients with locally advanced or metastatic sarcoma；Enrollment of 10 evaluable subjects in Phase I. If ≥2 subjects experience objective remission or SD lasting >12 weeks, proceed to Phase II to enroll an additional 20 evaluable subjects to further evaluation of the safety and efficacy of LTC004

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years；
2. Subjects with histologically or cytologically confirmed non-surgically treatable and failed standard therapy recommended by existing clinical standards of care or guidelines at screening (PD during treatment or PD after final treatment), or locally advanced or metastatic sarcoma that cannot tolerate standard therapy and/or for which there is currently no effective standard therapy (if recurrence or metastasis occurs during adjuvant therapy or within 6 months of completion, adjuvant therapy is considered a first-line treatment failure). Note: Embryonal rhabdomyosarcoma, follicular rhabdomyosarcoma, Ewing's sarcoma/primitive neuroectodermal tumor, gastrointestinal mesenchymal tumors, and malignant mesothelioma should be excluded.
3. At least one measurable tumor lesion based on RECIST V1.1 criteria；
4. ECOG PS ≤1；
5. Expected survival ≥12 weeks；
6. Adequate organ function；
7. Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for 6 months after the last infusion of LTC004.
8. Patients who have received any chemotherapy or anti-tumor monoclonal antibody drugs within 4 weeks prior to the first dose of study drug (excluding mitomycin and nitrosoureas within 6 weeks prior to the first dose of study drug）; small molecule targeted drugs within 2 weeks prior to the first dose of study drug; Chinese medicine therapy (Chinese medicine therapy with clear anti-tumor indications in the package insert ）within 4 weeks prior to the first dose of study drug；
9. Understands and provides written informed consent and willing to follow the requirements specified in protocol.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other mAbs.
2. Untreated, unstable or uncontrolled central nervous system (CNS) metastases with following exceptions:A. Clinically stable MRI scans and no progressive or uncontrolled neurologic symptoms or signs for at least 4 weeks prior to the first study treatment;
3. Patients with untreated or clinically symptomatic spinal cord compression that has not been controlled.
4. Patients with uncontrolled pleural effusion, pericardial effusion or abdominal effusion as judged by the investigator at screening;
5. Previous immunotherapy, including IL-2, IL-15, PD-1/L1 inhibitors, NK, and TCR-T cell therapy.
6. ≥2 malignant tumors within 5 years prior to first dose of drug；
7. Moderate to severe dyspnea at rest, severe primary lung disease, current need for continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonia due to advanced cancer or its complications; Grade ≥3 interstitial pneumonia during prior antineoplastic therapy；
8. Presence of severe infection within 4 weeks prior to first dose of medication，Presence of active infection requiring systemic antibiotic therapy with CTCAE grade ≥2 within 2 weeks prior to first dose
9. History of serious cardiovascular disease；
10. Active hepatitis B; hepatitis C infection; syphilis infection, active tuberculosis;
11. Patients with active, or previous autoimmune disease with potential for recurrence;
12. Immunodeficiency diseases or history of such diseases, including a positive serologic test for human immunodeficiency virus (HIV)
13. Arterial/venous thrombotic events within 6 months prior to the first dose of the drug;
14. Those who received radical radiation therapy within 4 weeks prior to the first dose and those who received palliative radiation within 14 days prior to the first dose.
15. Received other unlisted clinical investigational drug or treatment within 4 weeks prior to first dose.
16. Use of live or attenuated vaccines within 4 weeks prior to the first dose, or anticipated need for live or attenuated vaccines during the study period；
17. Major surgery (other than surgery for diagnostic purposes) within 4 weeks prior to the first dose, anticipation of major surgery (other than surgery for diagnostic purposes) during the study period, or diagnostic or low-invasive surgery within 7 days prior to the first dose (excluded for puncture biopsies).
18. Tumor invasion into peripheral vital organs (e.g., aorta and trachea) or risk of esophageal-tracheal fistula or esophageal-pleural fistula; history of gastrointestinal perforation and/or fistula within 6 months prior to the first dose of the drug；
19. Adverse effects of prior antitumor therapy have not recovered to CTCAE version 5.0 grade rating ≤1；
20. Patients who have received a previous allogeneic bone marrow/hematopoietic stem cell transplant or solid organ transplant；
21. Pregnant and lactating women；
22. Subjects who in the judgment of the investigator, have a history of other serious systemic disease or are unfit to participate in this trial for any other reason (the presence of psychiatric disorders in the patient that may affect compliance with the trial, alcohol, drug or substance abuse, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-26 (Estimated); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 12 months
  Antitumor efficacy of LTC004 treated sarcoma patients

SECONDARY OUTCOMES:
DOR | up to 12 months
  Duration of Response of LTC004 treated sarcoma patients
PFS rate | up to 12 months
  12 weeks and 24 weeks Progression-Free Survival rate of LTC004 treated sarcoma patients
OS | up to 12 months
  Overall Survival of LTC004 treated sarcoma patients

IPD SHARING:
Plan to Share IPD: No